CLINICAL TRIAL: NCT04484844
Title: Clinical Evaluation of Efficacy of Shield Force Plus Varnish Versus Sodium Fluoride on Cervical Dentin Hypersensitivity on Adult Patients: A Randomized Clinical Trial
Brief Title: Clinical Evaluation of Efficacy of Shield Force Plus Varnish VS Sodium Fluoride on Dentin Hypersensitivity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Feras Mustafa Fares Salem, Master's degree student - faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPER 20/7/2020
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Dentin Hypersensitivity; Dentin Desensitizing Agents
Keywords: Dentin hypersensitivity; Dentin sensitivity; Shield force plus; Dentin Desensitizing Agents; sodium fluoride varnish
MeSH Terms: conditions — Dentin Sensitivity | interventions — Tokuyama Shield Force Plus; Sodium Fluoride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Shield Force Plus Varnish (Experimental): Shield force plus (SFP), Self-reinforcing (SR) monomer technology supplied in the form of one component self-etching light-cured dental adhesive, which is characterized by an SR monomer component that penetrates the tooth substrate. Multi-point interactions with apatite calcium and three-dimensional cross-linking occur reactions.it forms a thin even, hard coating on the tooth surface that gives the tooth substrate a superior binding power.
  Interventions: Drug: TOKUYAMA SHIELD FORCE PLUS
- Sodium Fluoride varnish (Active Comparator): Topical application of varnish fluoride (sodium fluoride NaF) effect on exposed dentine as a desensitizing agent, the varnish fluoride process is caused by the reaction between NaF and calcium ions resulting in calcium fluoride crystals being deposited on the openings of the dentinal tubules that decrease pain.
  Interventions: Drug: Sodium Fluoride 5% Dental Varnish

INTERVENTIONS:
Drug: TOKUYAMA SHIELD FORCE PLUS — Self-reinforcing (SR) monomer technology
  Arms: Shield Force Plus Varnish
Drug: Sodium Fluoride 5% Dental Varnish — 5% NaF
  Arms: Sodium Fluoride varnish

SUMMARY:
The aim of the study to compare the clinical effectiveness of Shield Force Plus (SFP) versus sodium fluoride varnish in the management of hypersensitivity of cervical dentin in adult patients for 8weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good oral hygiene.
* The age range of 18-65 years.
* Patients from both gender.
* Patients suffering from pain due to dentin hypersensitivity.
* Patients with sound first upper molars.

Exclusion Criteria:

* Patients with teeth exhibiting mobility (grade 2 or 3).
* Patients with constant use of analgesic, carious lesions, fractured teeth, defective restorations or prosthesis.
* Patients with orthodontics appliance.
* Patients with allergy sufferers with any of the materials will be used in the study as shield force plus and sodium fluoride.
* Patients with carious, crowned upper first molars.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Dentin Hypersensitivity | Pre-intervention
  measurement of dentin hypersensitivity by VAS Scale
Dentin Hypersensitivity | 2 min
  measurement of dentin hypersensitivity by VAS Scale
Dentin Hypersensitivity | 1 week
  measurement of dentin hypersensitivity by VAS Scale
Dentin Hypersensitivity | 4 weeks
  measurement of dentin hypersensitivity by VAS Scale
Dentin Hypersensitivity | 8 weeks
  measurement of dentin hypersensitivity by VAS Scale

SECONDARY OUTCOMES:
Dentinal Tubule Occlusion | Pre-intervention
  percentage of dentinal tubule occlusion measure by scanning electron microscope SEM
Dentinal Tubule Occlusion | 8 weeks
  percentage of dentinal tubule occlusion measure by scanning electron microscope SEM